CLINICAL TRIAL: NCT06361225
Title: Routine Use of RUSH Protocol in the Intensive Care Unit- Does it Influence Patient Management? Prospective Observational Study
Brief Title: Routine Use of RUSH Protocol in the Intensive Care Unit
Status: Recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: 0075-24-MMC
Record Dates: First submitted 2024-03-31; First posted 2024-04-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: RUSH Protocol
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: evaluation with RUSH protocol — Daily evaluation of the patient via ultrasound using the RUSH protocol

SUMMARY:
The RUSH protocol has been used for several years for the rapid evaluation of a patient admitted to the emergency room with shock. Traditionally, its use was especially common in trauma victims, but later its use was extended to patients admitted to the emergency room with shock from any reason. The protocol includes rapid assessment with the guideness of ultrasound of heart contraction, assessment for pleural effusions, assessment of intra-abdominal blood (FAST), diagnosis of venous thrombosis (DVT), and rulling out hydronephrosis. It can also add a pupil size assessment and an evaluation of the gallbladder and bile ducts, as well as the size of the bladder. In intensive care, we use this protocol (or part of it) for the evaluation of a patient who is deteriorating in the ICU for an unknown reason . In some patients we use this protocol as a routine part of the physical examination as part of the daily patient evaluation.

We would like to investigate whether the routine use of the RUSH protocol as part of the daily patient evaluation in the general intensive care unit will lead to any change in the patient's management.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were admitted to the intensive care unit for any reason and were evaluated daily using the RUSH protocol.

Exclusion Criteria:Patients who were not evaluated using the RUSH protocol or for whom data were missing.

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were admitted to the intensive care unit for any reason and were evaluated daily using the RUSH protocol.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change of patient medical therapy | from day 0 to day 3 of performing the RUSH protocol
  Adding a new medical therapy= yes/no (1/0), changing the dose of an existing medical therapy (increase/decrease=1/0)
Performing unplanned laboratory tests | from day 0 to day 3 of performing the RUSH protocol
  Performing unplanned laboratory tests as a result of the RUSH protocol- yes/no (=1/0)
Performing unplanned image tests | from day 0 to day 3 of performing the RUSH protocol
  Performing unplanned image tests (CXR, CT etc.) as a result of the RUSH protocol- yes/no (=1/0)
Performing unplanned invasive procedure | from day 0 to day 3 of performing the RUSH protocol
  Performing unplanned invasive procedure (surgery, minimally invasive procedure)- yes/no (1/0)

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No